CLINICAL TRIAL: NCT07224360
Title: Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety of Anumigilimab (CSL324) in Adults With Sickle Cell Disease
Brief Title: Safety of Anumigilimab (CSL324) in Adults With Sickle Cell Disease (SCD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL324_2002; 2025-521154-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: Anemia; Genetic Disorder; Vaso-occlusive Crises
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Genetic Diseases, Inborn; Vaso-Occlusive Crises

STUDY DESIGN:
Intervention Model Description: This is a double blind, placebo controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anumigilimab (Experimental): Safety of Anumigilimab (CSL324) in Adults with Sickle Cell Disease (SCD)
  Interventions: Biological: Anumigilimab
- Placebo (Placebo Comparator): Participants will receive matching volume of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Anumigilimab — Participants will receive anumigilimab, escalated to a maximum dose guided by absolute neutrophil count (ANC) and safety concerns.
  Arms: Anumigilimab
Drug: Placebo — Volume matched saline will be administered SC.
  Arms: Placebo

SUMMARY:
This is a phase 2a, global, multicenter, randomized, double-blind, placebo-controlled study investigating the safety of anumigilimab administered subcutaneously (SC) at the maximum tolerated dose (MTD) in adult participants with SCD.

The primary aim of the study is to assess the safety of anumigilimab in participants with SCD. Participants will be treated for 64 weeks: for 12 weeks in the dose escalation period, where the dose will be escalated to each participant's individual MTD; and for 52 weeks at the MTD in the maintenance period.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged greater than or equal to (>=) 18 years on the day of signing the informed consent form.
* • Confirmed diagnosis of SCD of any genotype.
* • Experienced 1 to 12 VOCs requiring a visit to a medical facility and treatment with parenteral opioids or a parenteral nonsteroidal anti-inflammatory drug within the 12 months before Screening.
* • HU Regimen:
* a. On stable and well-tolerated Hydroxyurea (HU) regimen for at least 30 days before Screening.
* or
* b. HU was discontinued or refused (eg, due to concern of side effects or lack of effect).

Exclusion Criteria:

* • Absolute neutrophil count less than (<) 2.5 ×10^9 cells/Litre at Screening or Baseline (Week 1 Day 1).
* • If on SCD preventive medication, dose is not stable in the 30 days before Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2028-06-29 (Estimated); Study Completion 2028-06-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs), Overall and by severity, seriousness and relationship to Investigational Product (IP) | From baseline up to Week 75
Percentage of participants with TEAEs Overall and by severity, seriousness and relationship to IP | From baseline up to Week 75
Number of participants with Adverse Events of Special Interest (AESI) | From baseline up to Week 75
  The following AEs are to be reported as AESI: neutropenia (Common Terminology Criteria for Adverse Events [CTCAE] Grade 3 or 4), severe infection and neutropenic fever.
Percentage of participants with AESI | From baseline up to Week 75
  The following AEs are to be reported as AESI: neutropenia (CTCAE Grade 3 or 4), severe infection and neutropenic fever.
Number of participants with clinically relevant changes from baseline in laboratory assessments and vital signs | From baseline up to Week 75
Percentage of participants with clinically relevant changes from baseline in laboratory assessments and vital signs | From baseline up to Week 75

SECONDARY OUTCOMES:
Serum concentration of Anumigilimab | From the first dose of anumigilimab to Week 65
Annualized rate of Vaso-occlusive crisis (VOC) (medical facility) | During the maintenance period from Week 13 to Week 65
  VOC (medical facility) is defined as VOC that results in a visit to a medical facility and treatment with parenteral opioids or a parenteral nonsteroidal anti-inflammatory drug.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.